CLINICAL TRIAL: NCT01430949
Title: A Single-Arm Multi-Center Trial of Radiofrequency Ablation for the Treatment of Paroxysmal Atrial Fibrillation Using the Bard Over-the-Wire Ablation System
Brief Title: GENESIS Feasibility Study of the BARD Over-the-Wire Mesh Ablation System for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: GENESIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEP-4409-2010
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Catheter Ablation; Pulmonary Vein Isolation; Radio Frequency Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Over-the-Wire Mesh Ablation System (Experimental)
  Interventions: Procedure: Catheter Ablation of Paroxysmal Atrial Fibrillation

INTERVENTIONS:
Procedure: Catheter Ablation of Paroxysmal Atrial Fibrillation — Catheter ablation for the treatment of paroxysmal atrial fibrillation. A pulmonary vein isolation procedure will be performed using the OTW MAS and radiofrequency ablation.
  Other Names: GENESIS; BEP-4409; Bard Over-the-Wire Mesh Ablation System; OTW MAS; Paroxysmal Atrial Fibrillation; PAF; Feasibility

SUMMARY:
The Genesis Feasibility Study will collect clinical information on the use of the Bard Over-the-Wire Mesh Ablation System to access and perform electrophysiological mapping, cardiac stimulation and radiofrequency ablation in the region of the pulmonary vein (PV) ostia for the treatment of patients with Paroxysmal Atrial Fibrillation. Patients will be followed up for 12 months to assess the primary safety endpoint of Major Complications (a composite safety endpoint)and effectiveness, defined as Long-Term Success (freedom from recurrent atrial arrhythmia.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia seen by the physician. Its prevalence in the population increases with age, and it is estimated to affect over 4% of the population above the age of 60. Common approaches to AF management includes the use of anti-arrhythmic drugs to control the arrhythmia.

An alternative to treatment of AF using drug therapy is ablation of cardiac tissue, with the goal of disrupting the aberrant electrical pathways that cause AF through the creation of ablation lesions within the left atrium. There are several different approaches to creating lesions to treat AF, although both substrate derived and focal AF mechanisms share a common ablation therapy protocol in which the PVs are isolated by a series of ablation lines placed endocardially, either around the PV ostia or more proximally from the PV ostia at the atrial carinae.

The Over-the-Wire Mesh Ablation System (OTW MAS) catheter is a combined mapping and ablation catheter designed to create lesions at the PV ostium. The Genesis Feasibility Study is designed to collect clinical information on the use of the OTW MAS to access and perform electrophysiological mapping, cardiac stimulation and radiofrequency ablation in the region of the pulmonary vein (PV) ostia for the treatment of patients with Paroxysmal Atrial Fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic PAF refractory to at least one Class I-IV antiarrhythmic drug.
* Minimum one documented PAF episode >30 sec duration within prior 12 months.
* Minimum three PAF episodes during prior 12 months.
* 18 years or older.

Exclusion Criteria:

* AF due to reversible causes.
* More than 2 cardioversions during the 6 months
* Previous surgical or catheter based ablation of the LA to treat AF.
* Permanent or persistent AF.
* Requirement for ablation lesions other than those defined in protocol
* LA > 50 mm in major dimension(measured by TTE).
* Any single PV > 25 mm in major diameter and/or presence of common os not suitable for ablation
* Ejection fraction <35%.
* Patent foramen ovale (PFO)or atrial septal defect (ASD)
* Cardiac myopathy (e.g., HOCM, cardiac sarcoidosis).
* Myocardial infarction in previous 2 months screening.
* Currently unstable angina.
* Any cardiac surgery in previous 3 months prior to screening.
* Implantable device capable of recording cardiac rhythm, (e.g ICD, pacemaker or implantable loop recorder.
* Clinically significant valvular heart disease or a replacement heart valve.
* Congestive heart failure (NYHA classification III or IV).
* Renal dialysis or creatinine > 2.0 mg/dl.
* Contraindication to anti-coagulation therapy (e.g., warfarin, heparin).
* Contraindication to transseptal procedure.
* Any cerebral ischemic event, including TIA in the 6 months prior to screening.
* Any known uncontrolled bleeding or thrombotic disorder.
* Women who are known to be pregnant or nursing.
* Uncontrolled hyperthyroidism.
* Patients currently enrolled in any other study during the 30 days prior to screening.
* Any other significant uncontrolled or unstable medical condition (e.g., active systemic infection).
* A life expectancy of less than one year.
* Currently documented intracardiac thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 months
  Freedom from recurrence of symptomatic atrial fibrillation, atrial tachycardia or atrial flutter. Includes both acute success (successful electrical isolation of all pulmonary veins) and chronic success. Re-treatment for AF with ablation during the 3 month blanking period will not constitute a treatment failure.

SECONDARY OUTCOMES:
Safety | 12 months
  Incidence of device-related early-onset primary serious adverse events or adverse device effects. Includes serious adverse events occurring within 7 days of the index procedure and diagnosed at any time during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: David Ciavarella, MD, Study Chair — CR Bard Inc
Locations (6):
- Canada (2):
  - University Hospital, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
- Germany (3):
  - Herz-und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Deutsches Herzzentrum Berlin (DHZB), Berlin
  - Herzzentrum Mūnchen, Munich
- The Heart Hospital, London, United Kingdom